CLINICAL TRIAL: NCT06540248
Title: Real-life Clinical Experience With a Minimally Invasive Syringe Adapter for Catheter Free Instillation of Intravesical Treatments
Brief Title: Real-life Clinical Experience With Ialuadapter Study
Acronym: Ialuadapter
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Dick Janssen, MD PhD, Radboud University Medical Center
Other Study IDs: Ialudapter Study
Record Dates: First submitted 2024-07-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Interstitial Cystitis, Chronic; Overactive Bladder Syndrome; Recurrent Urinary Tract Infection
Keywords: IALUDAPTER; intravesical therapy; GAG therapy; Intravesical treatment; IC/BPS; recurrent urine tract infection; catheterization
MeSH Terms: conditions — Cystitis, Interstitial; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 61 patients evaluated: with IC/BPS (n=48), rUTI (n=6) and mixed /other diagnoses (including OAB; n= 7)
  Interventions: Device: Ialuadapter

INTERVENTIONS:
Device: Ialuadapter — minimally invasive syringe device for bladder catherization

SUMMARY:
A retrospective study from a single center was performed. Quantitative and qualitative data was obtained on the use of the syringe adapter (IALUADAPTER®) in 61 patients with IC/BPS (n=48), rUTI (n=6) and mixed /other diagnoses (including OAB; n= 7) who were receiving intravesical therapy. The evaluation period was 6 months during 2018-2019. Reasons for trying the syringe adapter, reasons for continuing with it and occurrence of UTIs before and during the evaluation period were recorded. In addition, 3 year follow-up data were obtained to assess long-term usage of the syringe adapter.

DETAILED DESCRIPTION:
Introduction Intravesical treatment is currently dependent on catheterization which can cause urethral discomfort and risk of urinary tract infections in selected patient groups such as interstitial cystitis / bladder pain syndrome (IC/BPS), overactive bladder syndrome (OAB) and recurrent urinary tract infections (rUTI). This study describes real-life clinical experience of a minimally invasive syringe adapter (Ialudapter®) for catheter-free instillation of intravesical treatment.

Methods A retrospective study from a single center was performed. Quantitative and qualitative data was obtained on the use of the syringe adapter (IALUADAPTER®) in 61 patients with IC/BPS (n=48), rUTI (n=6) and mixed /other diagnoses (including OAB; n= 7) who were receiving intravesical therapy. The evaluation period was 6 months during 2018-2019. Reasons for trying the syringe adapter, reasons for continuing with it and occurrence of UTIs before and during the evaluation period were recorded. In addition, 3 year follow-up data were obtained to assess long-term usage of the syringe adapter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IC/BPS, recurrent UTIs and/or OAB
* Receiving intravesical instillations with a conventional single-use catheter before the syringe adapter evaluation period which took place between September 2018 and the end of February 2019 (6m).

Exclusion Criteria:

* Patients with a high post-void residue of >100ml or with an indwelling catheter were excluded from the analyses.
* Patients who cannot sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with IC/BPS, recurrent UTIs and/or OAB
  * Receiving intravesical instillations with a conventional single-use catheter before the syringe adapter evaluation period which took place between September 2018 and the end of February 2019 (6m).
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who reported success (in using syringe adapter) Yes/No | 6 months
  pt self reported general assessment of successful instillation using the syringe adapter

SECONDARY OUTCOMES:
PRO; patient reported reasons for trying syringe adapter in stead of regular catheter (5 options) | 6 months
  patient reported subjective reasons for trying the syringe adapter: options: urethral pain, convenience, fear of catheter, urine tract infections or other
Total number of UTI's during syringe adapter use amongst all patients | 6 months
  Recorded UTI's reported in electronic patient database during the time they used syringe adapter
Number of participants who use syringe adapter 3 years after initial assessment (yes/no) | 1 yr
  long term adherence to syringe adapter (still using in in clinical practice)
PRO ; patient reported reasons to continue syringe adapter (5 options) | 6 months
  Subjective reasons given by patients for continuing with syringe adapter compared to regular catheter. Option were : hope for fewer urine tract infections, less pain, easier to use, self -sustainability, other)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided